CLINICAL TRIAL: NCT06528899
Title: Physiotherapy in Emergency Department: a Service Analysis From a French Hospital
Status: Completed | Type: Observational
Sponsor: Université de Nantes (Other)
Responsible Party: Principal Investigator, Guillaume Le Sant, PT, PhD - Researcher, Université de Nantes
Other Study IDs: KiUrge-retro
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Fall Patients; Pain; Sprains; Respiratory Insufficiency; Vertigo; Illness Behavior
Keywords: physical therapy; patient pathway; patient care management
MeSH Terms: conditions — Pain; Sprains and Strains; Respiratory Insufficiency; Vertigo; Illness Behavior | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency Physiotherapy (E-PT): Subcohort of patients receiving a referral + Emergency Physiotherapy (E-PT) during their visit to Emergency Department
  Interventions: Behavioral: Physical Therapy
- control (CTL): Subcohort of patients receiving a referral + but no Emergency Physiotherapy (E-PT) during their visit to Emergency Department

INTERVENTIONS:
Behavioral: Physical Therapy — Assessment and/or treatment by physitoherapist during the visit
  Groups: Emergency Physiotherapy (E-PT)

SUMMARY:
The skills of physiotherapists have been employed to enhance access to optimal care in Emergency Departments (ED). No study has yet been conducted on the practices in France. The primary objective of this study was to describe the French practices of physiotherapy within an ED, and to secondary examine the effect on patient discharge.

DETAILED DESCRIPTION:
A retrospective observational study was conducted on patients who received a referral for physiotherapy in the ED (E-PT) of the Universitarian Hospital of Nantes during a six-month observation period in 2022. A total of 461 medical records were extracted, including patient characteristics and the main chief complaint at the time of admission. Details on the delivery of E-PT were collected, as well as the end status at the exit of the ED. Descriptive statistics were performed to analyse the data. A propensity score analysis examined the association between the patients' status at the exit of the ED and E-PT.

ELIGIBILITY:
Inclusion Criteria:

* admission in the Emergency Departement
* aged over 18
* refferal for physiotherapy within the Emergency Department

Exclusion Criteria:

* death
* no admission within the Emergency Department (only administrative purposes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients visiting the Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Discharge at the exit of ED | up to 7 days (date of exit)
  the type of discharge (home / hospitalisation)

SECONDARY OUTCOMES:
Length of stay | up to 7 days (date of exit)
  duration of stay in the ED

OTHER OUTCOMES:
Age | date of presenting to ED
  Age of patients
Day of admission | date of presenting to ED
  day of the week
Chief complaint | date of presenting to ED
  The chief complaint for visiting the ED
Gender | date of presenting to ED
  gender of patients
Unit of referral | date of presenting to ED
  the unit of medical referral for E-PT

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Le Sant, PhD, Principal Investigator — guillaume.le-sant@univ-nantes.fr
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - Université de Nantes - MIP UR 4334 (Motricity, Movement, Interactions), Nantes

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author, [GLS], upon reasonable request. The data is not publicly available or to reusable due to privacy and ethical restrictions.